CLINICAL TRIAL: NCT00684060
Title: A Phase II, Randomized, Controlled, Double-Blind Pilot Trial Evaluating the Safety and Effect of Administration of Bone Marrow Mononuclear Cells Two to Three Weeks Following Acute Myocardial Infarction
Brief Title: Use of Adult Autologous Stem Cells in Treating People 2 to 3 Weeks After Having a Heart Attack (The Late TIME Study)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Dr Lemuel A Moye III, Professor - School of Public Health, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 578; 1U01HL087318 (NIH); 1 U01-HL-087318-01 (Project 2)
Record Dates: First submitted 2008-05-22; First posted 2008-05-26 (Estimated); Results first posted 2012-05-04 (Estimated); Last update posted 2015-07-10 (Estimated); Status verified 2015-07

CONDITIONS: Left Ventricular Dysfunction
Keywords: Acute Myocardial Infarction; Global Left Ventricular Ejection Fraction; Regional Left Ventricular Ejection Fraction; Left Ventricular Mass; Infarct Size; End Systolic Volume; End Diastolic Volume
MeSH Terms: conditions — Ventricular Dysfunction, Left | interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive active stem cell infusion 2 to 3 weeks after a percutaneous coronary intervention (PCI).
  Interventions: Biological: Adult stem cells
- 2 (Placebo Comparator): Participants will receive placebo infusion (5% human serum albumin [HSA]) 2 to 3 weeks after a PCI.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Adult stem cells — One time infusion of approximately 150 million total nucleated cells (TNC) in 30 ml of 5% HSA/saline solution
  Other Names: Adult autologous stem cells; Bone marrow mononucleated cells
  Arms: 1
Biological: Placebo — One time infusion of 30 ml of HSA (5%)
  Other Names: Human serum albumin; HSA
  Arms: 2

SUMMARY:
More than 1 million Americans suffer heart attacks each year. Although current treatments are able to stabilize the condition of the heart, none is able to restore heart function as it was prior to the heart attack. Adult stem cells, which are immature cells that can become many different types of cells, may offer a potential means of reversing or preventing permanent damage caused by a heart attack. Recent studies have shown promise in using adult stem cells from bone marrow to reverse damage to the heart muscle caused by a heart attack, but more research is needed to assess the safety and effectiveness of stem cell use and to discover the best time to administer treatment. This study will evaluate the safety and effectiveness of using adult stem cell infusions 2 to 3 weeks after a heart attack for improving heart function in people who have had a recent heart attack and a common procedure called a percutaneous coronary intervention (PCI).

DETAILED DESCRIPTION:
Heart attacks are a leading cause of death for both men and women in the United States. A heart attack occurs when blood flow to the heart is restricted, commonly due to a blood clot that has formed in one of the coronary arteries. If the clot becomes large enough, blood flow to the heart can be blocked almost completely and the heart muscle in that area can suffer permanent injury or death. Although a PCI can be used to open up the blocked artery and restore blood flow to the heart muscle, there may be a significant amount of heart tissue that has been irreversibly damaged. Recent studies have shown that adult stem cells from bone marrow may be able to improve heart function after a heart attack. These specialized cells may have the ability to promote blood vessel growth, prevent cell death, and transform themselves into a number of tissues, including muscle. After an acute heart attack, a remodeling process is initiated in the heart in an attempt to compensate for damaged areas. Consequently, the condition of the heart muscle several weeks after a heart attack may differ considerably from the heart's condition during the acute setting. For some patients, delaying the delivery of the stem cells until 2 to 3 weeks after a heart attack may be better than initiating treatment during the acute phase. This study will evaluate the safety and effectiveness of placing adult stem cells into injured heart muscle 2 to 3 weeks after a heart attack for improving heart function in people who have had a recent heart attack and a PCI.

Participation in this study will last 24 months. All participants will first undergo baseline assessments that will include a medical history, a physical exam, an electrocardiogram (ECG), blood draws, an echocardiogram, and a magnetic resonance imaging (MRI) test. Participants will then be assigned randomly to receive stem cells or placebo between 2 and 3 weeks after their heart attack. The morning of the stem cell or placebo infusion, participants will undergo a blood draw and a bone marrow aspiration procedure of the hip bone to collect the stem cells. Later the same day, either stem cells or placebo will be infused through a catheter and into the damaged area of the heart.

For the first 24 hours after the infusion, participants will be asked to wear a small ECG machine called a Holter monitor. Participants will also be asked to record their temperature twice a day for a month after the infusion. Participants will return for follow-up visits at Months 1, 3, 6, 12, and 24 and will repeat many of the baseline assessments.

ELIGIBILITY:
Inclusion criteria

1. Patients at least 21 years of age.
2. Patients with first acute MI and subsequent successful primary percutaneous coronary intervention (PCI) in an artery at least 2.5 mm in diameter occurring two to three weeks before recruitment.
3. No contraindications to undergoing cell therapy procedure within two to three weeks following AMI and PCI.
4. Hemodynamic stability as defined as no requirement for IABP, inotropic or blood pressure supporting medications.
5. Ejection fraction following reperfusion with PCI <=45% as assessed by echocardiography.
6. Consent to protocol and agree to comply with all follow-up visits and studies.
7. Women of child bearing potential willing to use an active form of birth control.

Exclusion criteria

Patients will be excluded from the study if they meet any of the following conditions:

1. History of sustained ventricular arrhythmias not related to their AMI (evidenced by previous holter monitoring and/or medication history for sustained ventricular arrhythmias in patient's medical chart).
2. Require CABG or PCI due to the presence of residual coronary stenosis >70% luminal obstruction in the non-infarct related vessel (Additional PCI of non-culprit vessels may be performed prior to enrollment).
3. History of any malignancy within the past five years excluding non-melanoma skin cancer or cervical cancer in-situ.
4. History of chronic anemia (hemoglobin (Hb) <9.0 mg/dl).
5. History of thrombocytosis (platelets >500k).
6. History of thrombocytopenia in the absence of recent evidence that platelet counts are normal
7. Known history of elevated INR (PT) or PTT.
8. Life expectancy less than one year.
9. History of untreated alcohol or drug abuse.
10. Currently enrolled in another Investigational drug or device trial
11. Previous CABG.
12. Previous MI resulting in LV dysfunction (LVEF <55%)
13. History of stroke or transient ischemic attack (TIA) within the past six months.
14. History of severe valvular heart disease (aortic valve area <1.0 cm2 or >3+ mitral regurgitation).
15. Pregnancy or breast feeding
16. Subjects with a known history of HIV, or has active hepatitis B, active hepatitis C, or active tuberculosis (TB)
17. Patients with active inflammatory or autoimmune disease on chronic immunosuppressive therapy.
18. Contraindications to cMRI.
19. Previous radiation to the pelvis with white blood cell count (WBC) and platelet counts below hospital specific normal values.
20. Women child bearing potential not willing to practice an active form of birth control.
21. Chronic liver disease that might interfere with survival or treatment with cell therapy.
22. Chronic renal insufficiency as defined by a creatinine ≥2.0 mg/dL or requires chronic dialysis.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Actual)
Dates: Start 2008-07; Primary Completion 2011-08 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Simari, MD, Study Chair — Cardiovascular Cell Therapy Research Network
Locations (5):
- United States (5):
  - University of Florida - Department of Medicine, Gainesville, Florida
  - Minneapolis Heart Institute Foundation, Minneapolis, Minnesota
  - Cleveland Clinic, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Texas Heart Institute, Houston, Texas

REFERENCES:
- [Background] Traverse JH, Henry TD, Vaughan DE, Ellis SG, Pepine CJ, Willerson JT, Zhao DX, Simpson LM, Penn MS, Byrne BJ, Perin EC, Gee AP, Hatzopoulos AK, McKenna DH, Forder JR, Taylor DA, Cogle CR, Baraniuk S, Olson RE, Jorgenson BC, Sayre SL, Vojvodic RW, Gordon DJ, Skarlatos SI, Moye LA, Simari RD; Cardiovascular Cell Therapy Research Network. LateTIME: a phase-II, randomized, double-blinded, placebo-controlled, pilot trial evaluating the safety and effect of administration of bone marrow mononuclear cells 2 to 3 weeks after acute myocardial infarction. Tex Heart Inst J. 2010;37(4):412-20. PMID 20844613
- [Background] Gee AP, Richman S, Durett A, McKenna D, Traverse J, Henry T, Fisk D, Pepine C, Bloom J, Willerson J, Prater K, Zhao D, Koc JR, Ellis S, Taylor D, Cogle C, Moye L, Simari R, Skarlatos S. Multicenter cell processing for cardiovascular regenerative medicine applications: the Cardiovascular Cell Therapy Research Network (CCTRN) experience. Cytotherapy. 2010 Sep;12(5):684-91. doi: 10.3109/14653249.2010.487900. PMID 20524773
- [Background] Zierold C, Carlson MA, Obodo UC, Wise E, Piazza VA, Meeks MW, Vojvodic RW, Baraniuk S, Henry TD, Gee AP, Ellis SG, Moye LA, Pepine CJ, Cogle CR, Taylor DA. Developing mechanistic insights into cardiovascular cell therapy: Cardiovascular Cell Therapy Research Network Biorepository Core Laboratory rationale. Am Heart J. 2011 Dec;162(6):973-80. doi: 10.1016/j.ahj.2011.05.024. PMID 22137069
- [Result] Traverse JH, Henry TD, Ellis SG, Pepine CJ, Willerson JT, Zhao DX, Forder JR, Byrne BJ, Hatzopoulos AK, Penn MS, Perin EC, Baran KW, Chambers J, Lambert C, Raveendran G, Simon DI, Vaughan DE, Simpson LM, Gee AP, Taylor DA, Cogle CR, Thomas JD, Silva GV, Jorgenson BC, Olson RE, Bowman S, Francescon J, Geither C, Handberg E, Smith DX, Baraniuk S, Piller LB, Loghin C, Aguilar D, Richman S, Zierold C, Bettencourt J, Sayre SL, Vojvodic RW, Skarlatos SI, Gordon DJ, Ebert RF, Kwak M, Moye LA, Simari RD; Cardiovascular Cell Therapy ResearchNetwork. Effect of intracoronary delivery of autologous bone marrow mononuclear cells 2 to 3 weeks following acute myocardial infarction on left ventricular function: the LateTIME randomized trial. JAMA. 2011 Nov 16;306(19):2110-9. doi: 10.1001/jama.2011.1670. Epub 2011 Nov 14. PMID 22084195
- [Derived] Shahrivari M, Wise E, Resende M, Shuster JJ, Zhang J, Bolli R, Cooke JP, Hare JM, Henry TD, Khan A, Taylor DA, Traverse JH, Yang PC, Pepine CJ, Cogle CR; Cardiovascular Cell Therapy Research Network (CCTRN). Peripheral Blood Cytokine Levels After Acute Myocardial Infarction: IL-1beta- and IL-6-Related Impairment of Bone Marrow Function. Circ Res. 2017 Jun 9;120(12):1947-1957. doi: 10.1161/CIRCRESAHA.116.309947. Epub 2017 May 10. PMID 28490433
- [Derived] Bhatnagar A, Bolli R, Johnstone BH, Traverse JH, Henry TD, Pepine CJ, Willerson JT, Perin EC, Ellis SG, Zhao DX, Yang PC, Cooke JP, Schutt RC, Trachtenberg BH, Orozco A, Resende M, Ebert RF, Sayre SL, Simari RD, Moye L, Cogle CR, Taylor DA; Cardiovascular Cell Therapy Research Network (CCTRN). Bone marrow cell characteristics associated with patient profile and cardiac performance outcomes in the LateTIME-Cardiovascular Cell Therapy Research Network (CCTRN) trial. Am Heart J. 2016 Sep;179:142-50. doi: 10.1016/j.ahj.2016.06.018. Epub 2016 Jul 6. PMID 27595689
- [Derived] Cogle CR, Wise E, Meacham AM, Zierold C, Traverse JH, Henry TD, Perin EC, Willerson JT, Ellis SG, Carlson M, Zhao DX, Bolli R, Cooke JP, Anwaruddin S, Bhatnagar A, da Graca Cabreira-Hansen M, Grant MB, Lai D, Moye L, Ebert RF, Olson RE, Sayre SL, Schulman IH, Bosse RC, Scott EW, Simari RD, Pepine CJ, Taylor DA; Cardiovascular Cell Therapy Research Network (CCTRN). Detailed analysis of bone marrow from patients with ischemic heart disease and left ventricular dysfunction: BM CD34, CD11b, and clonogenic capacity as biomarkers for clinical outcomes. Circ Res. 2014 Oct 24;115(10):867-74. doi: 10.1161/CIRCRESAHA.115.304353. Epub 2014 Aug 18. PMID 25136078
- See also: Click here for more information on this study at the Cardiovascular Cell Therapy Research Network (CCTRN) — http://www.cctrn.org
- See also: Click here for the National Heart, Lung, and Blood Institute — http://www.nhlbi.nih.gov/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment took place at five Network centers and their associated satellite facilities between July 8, 2008 and February 28, 2011. The main centers are located in Ohio, Texas, Florida, Minnesota, and Tennessee. Study brochures, patient informational DVDs, and clinical trials.gov were among the tools used for recruitment.
Groups:
- Stem Cell Arm: Participants will receive active stem cell infusion 2 to 3 weeks after a percutaneous coronary intervention (PCI).
- Placebo Arm: Participants will receive placebo infusion (5% human serum albumin [HSA]) 2 to 3 weeks after a PCI.
Period: Overall Study
Arm/Group | Stem Cell Arm | Placebo Arm
Started | 58 | 29
Completed | 55 | 26
Not Completed | 3 | 3
Not completed — Lost to Follow-up | 1 | 0
Not completed — New stenosis identified | 1 | 0
Not completed — Unable to collect MRI | 1 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stem Cell Arm | Placebo Arm | Total
Number analyzed (Participants) | 58 | 29 | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.6 (11) | 54.6 (11) | 57 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 15
  Male | 46 | 26 | 72
Region of Enrollment [Number; unit: participants]
  United States | 58 | 29 | 87

OUTCOME MEASURES:

1. Primary Outcome: Global Left Ventricular Function
Description: Left ventricular ejection fraction (global) as assessed via cardiac MRI. Values reported represent the change in Global EF from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in Global EF from baseline to six months.
Measure: Mean (Standard Deviation); unit: percentage of ejection fraction
Arm/Group | Stem Cell Arm | Placebo Arm
Number analyzed (Participants) | 55 | 26
percentage of ejection fraction | 0.5 (8.2) | 3.6 (9.3)
Statistical Analysis 1: Comparison: Stem Cell Arm vs Placebo Arm; Comparison of change in global LVEF in the active group minus change in global LVEF in the control group. 80 percent power based on BOOST results; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Threshold 0.05; No adjustment for multiple comparisons; Mean Difference (Net) = -3.0, 95% CI 2-sided [-7.05 to .95], Standard Error of Mean 8.6

2. Secondary Outcome: Combined Endpoint
Description: Combined endpoint: first of death, reinfarction, repeat revascularization, and hospitalization for heart failure. This is measured as the number of events by treatment group over the 6 month follow up period.
Time Frame: Measured at Baseline and Month 6
Population: All randomized patients were followed for clinical outcomes. However the paucity of events precluded a reliable time to event analysis.
Measure: Number; unit: events
Arm/Group | Stem Cell Arm | Placebo Arm
Number analyzed (Participants) | 58 | 29
events | 3 | 4
Statistical Analysis 1: Comparison: Stem Cell Arm vs Placebo Arm; comparison of the proportion of events in patients in the active group to those in patients in the control group; Test type: Superiority or Other; p < 0.05, Fisher Exact; Odds Ratio (OR) = 0.30, 95% CI [0.08 to 1.17]

3. Secondary Outcome: Left Ventricular Mass
Description: Left ventricular mass (LV mass. Values reported represent the change in LV mass from baseline to six months.)
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in LV mass from baseline to six months.
Measure: Mean (Standard Deviation); unit: g
Arm/Group | Stem Cell Arm | Placebo Arm
Number analyzed (Participants) | 55 | 26
g | -12.0 (18.1) | -10.8 (15.2)
Statistical Analysis 1: Comparison: Stem Cell Arm vs Placebo Arm; Comparison of change in the active group minus change in global LVEF in the control group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = -1.2, 95% CI 2-sided [-9.3 to 6.8], Standard Error of Mean 17.2

4. Secondary Outcome: End Diastolic Volume Index
Description: Left ventricular end diastolic volume index. Values reported represent the change in LV end diastolic index from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in LV end diastolic index from baseline to six months.
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Stem Cell Arm | Placebo Arm
Number analyzed (Participants) | 55 | 26
mL/m2 | 3.4 (23.4) | 2.7 (18.1)
Statistical Analysis 1: Comparison: Stem Cell Arm vs Placebo Arm; Comparison of change in the active group minus change in global LVEF in the control group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 0.7, 95% CI 2-sided [-9.5 to 10.9], Standard Error of Mean 21.8

5. Secondary Outcome: End Systolic Volume Index
Description: Left ventricular end systolic volume index. Values reported represent the change in LV end systolic volume index from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in LV end systolic volume index from baseline to six months.
Measure: Mean (Standard Deviation); unit: mL/m2
Arm/Group | Stem Cell Arm | Placebo Arm
Number analyzed (Participants) | 55 | 26
mL/m2 | 0.2 (14.0) | -2.3 (14.7)
Statistical Analysis 1: Comparison: Stem Cell Arm vs Placebo Arm; Comparison of change in the active group minus change in the control group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = 2.5, 95% CI 2-sided [-4.1 to 9.2], Standard Error of Mean 14.2

6. Secondary Outcome: Infarct Volume
Description: Infarct volume(mL). Values reported represent the change in infarct volume from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included.
  Values reported represent the change in infarct volume from baseline to six months.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Stem Cell Arm | Placebo Arm
Number analyzed (Participants) | 55 | 25
mL | -3.5 (19.0) | -2.0 (14.4)
Statistical Analysis 1: Comparison: Stem Cell Arm vs Placebo Arm; Comparison of change in the active group minus change in the control group; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = -1.5, 95% CI [-9.9 to 6.9], Standard Error of Mean 17.7

7. Primary Outcome: Regional Left Ventricular Function (Infarct Zone Wall Motion)
Description: One of two calculated values of regional left ventricular function as assessed via cardiac MRI. The infarct zone is defined as the cMRI segments with the largest 2 signal intensity enhancement measures with gadolinium (using a 17-segment model).Values reported represent the change in wall motion over time in the infarct zone from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Only participants with both baseline and 6 month MRI images available are included. One patient was excluded from the analysis due to incomplete signal intensity enhancement data.
  Values reported represent the change in wall motion over time in the infarct zone from baseline to six months.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stem Cell Arm | Placebo Arm
Number analyzed (Participants) | 55 | 25
mm | 0.3 (4.3) | 1.0 (4.5)
Statistical Analysis 1: Comparison: Stem Cell Arm vs Placebo Arm; Comparison of change in infarct zone wall motion in the active group minus change in global LVEF in the control group. 80 percent power based on BOOST results; Test type: Superiority or Other; p < 0.05, t-test, 2 sided — Unadjusted; Mean Difference (Net) = -0.7, 95% CI 2-sided [-2.8 to 1.3], Standard Error of Mean 4.4

8. Primary Outcome: Regional Left Ventricular Function (Border Zone Wall Motion)
Description: Two of two calculated values of regional left ventricular function assessed via cardiac MRI. The border zone is defined as those regions adjacent to the infarct zone in which the cMRI signal intensity enhancement were in the 10%-75% range. Values reported represent the change in wall motion over time in the border zone of the infarct from baseline to six months.
Time Frame: Measured at Baseline and Month 6
Population: Five patients were excluded from analysis due to incomplete signal intensity enhancement data (1) or lack of a signal intensity enhancement signal in the border zone (4).
  Values reported represent the change in wall motion over time in the border zone of the infarct from baseline to six months.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Stem Cell Arm | Placebo Arm
Number analyzed (Participants) | 53 | 23
mm | 0.5 (7.2) | 3.2 (6.3)
Statistical Analysis 1: Comparison: Stem Cell Arm vs Placebo Arm; Comparison of change in border zone wall motion in the active group minus change in global LVEF in the control group. 80 percent power based on BOOST results; Test type: Superiority or Other; p < 0.05, t-test, 2 sided; Mean Difference (Net) = -2.6, 95% CI [-6.0 to 0.8], Standard Error of Mean 6.9

ADVERSE EVENTS:
Time Frame: Events reported are from Randomization Date to the 6 month endpoint data collection window (i.e. 210 days post intervention)
Arm/Group | Stem Cell Arm | Placebo Arm
Serious Adverse Events (participants affected / at risk) | 8/58 | 14/29
Other Adverse Events (participants affected / at risk) | 13/58 | 14/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Arm (N=58) | Placebo Arm (N=29)
Chest Pain (Cardiac disorders) | 6 (9) | 8 (8)
Heart Failure (Cardiac disorders) | 2 (2) | 2 (2)
Left Ventricular Thrombus (Cardiac disorders) | 0 (0) | 2 (2)
Tachycardia (Cardiac disorders) | 0 (0) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Arm (N=58) | Placebo Arm (N=29)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Chest Pain (Cardiac disorders) | 4 (5) | 4 (4)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 4 (4) | 2 (2)
Syncope (Cardiac disorders) | 1 (1) | 2 (2)

LIMITATIONS AND CAVEATS:
Lack of in-vivo testing of cell product. While there are several different approaches to measure myocardial strain (myocardial tagging, DENSE, etc.), these were not employed in this study due to the need for specialized expertise at each site.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes